CLINICAL TRIAL: NCT06921681
Title: Transbronchial EBUS-guided TBNA and Cryobiopsy of Mediastinal Lymph Nodes in Patients Nonsuspicious for Lung Cancer, Using Different Cryoprobe Freezing Times
Brief Title: Ultrasound-guided Cryobiopsy of Mediastinal/Hilar Lymph Nodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Aarau Cantonal Hospital (KSA) (Unknown); Waid City Hospital, Zurich (Other); Kantonsspital Winterthur KSW (Other); Unispital Basel (Unknown); Spital Uster AG, Uster, Switzerland (Unknown); Clinique des Grangettes, Chêne-Bougeries (Unknown); Insel Gruppe AG, University Hospital Bern (Other); Réseau Hospitalier Neuchâtelois (Other); University of Lausanne Hospitals (Other); Cantonal Hospital of St. Gallen (Other); Ospedale Regionale Bellinzona e Valli (Other); HUG - Hôpitaux universitaires de Genève (Unknown); Kantonsspital Chur, Switzerland (Unknown); Hôpital du Valais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-00885
Record Dates: First submitted 2025-03-10; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer (NSCLC)
Keywords: EBUS; Cryobiopsy; TBNA; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 6 sec (Active Comparator): EBUS-guided CBs of mediastinal/hilar lymph nodes will be done with 6 seconds of cryoprobe freezing time ("group 6sec.") before the biopsy together with the whole EBUS bronchoscope is extracted.
  Interventions: Device: Cryobiopsy of lymph nodes group 6 sec
- group 3 sec (Active Comparator): EBUS-guided CBs of mediastinal/hilar lymph nodes will be done with 3 seconds of cryoprobe freezing time ("group 3sec.") before the biopsy together with the whole EBUS bronchoscope is extracted.
  Interventions: Device: Cryobiopsy lymphnode group 3 sec

INTERVENTIONS:
Device: Cryobiopsy of lymph nodes group 6 sec — Included patients receive transbronchial access with EBUS needle (19, 21 or 22 gauge needle) Hereafter, three times EBUS-TBNA followed by four EBUS-guided-CBs with a 1.1mm cryoprobe will be performed. Included patients are 1:1 randomized to receive CB with cryoprobe activated for either 3 sec of freezing time (group "3sec") or 6 sec. of freezing time (group "6sec") before the biopsy together with the whole EBUS bronchoscope is extracted. The EBUS-guided CB will be conducted four times in each group. Aiming access to one lymph node if one lymph node cannot be punctured, another lymph node will be chosen. Even if tissue-extraction out of a lymph node via cryoprobe fails once to several times, overall no more than 4 attempts for cryobiopsy will be done
  Arms: group 6 sec
Device: Cryobiopsy lymphnode group 3 sec — Included patients receive transbronchial access with EBUS needle (19, 21 or 22 gauge needle) Hereafter, three times EBUS-TBNA followed by four EBUS-guided-CBs with a 1.1mm cryoprobe will be performed. Included patients are 1:1 randomized to receive CB with cryoprobe activated for either 3 sec of freezing time (group "3sec") or 6 sec. of freezing time (group "6sec") before the biopsy together with the whole EBUS bronchoscope is extracted. The EBUS-guided CB will be conducted four times in each group. Aiming access to one lymph node if one lymph node cannot be punctured, another lymph node will be chosen. Even if tissue-extraction out of a lymph node via cryoprobe fails once to several times, overall no more than 4 attempts for cryobiopsy will be done
  Arms: group 3 sec

SUMMARY:
EBUS-guided cryobiopsy of mediastinal and hilar lymph nodes has shown to be a useful diagnostic tool to obtain tissue for histological analysis and further targeted therapies in lung malignancies. Due to the large size and better quality of the tissue samples, a higher diagnostic yield than with transbronchial needle aspiration (TBNA) can be expected, especially in non-solid tumors. In previous studies different biopsy protocols were used. The freezing time of cryoprobe (which defines the sample sizes) ranged from 3 to 7 s and the number of biopsies was between 1 and 4 samples. It is therefore unclear what freezing times and biopsy frequency are required to obtain the best histological information.

DETAILED DESCRIPTION:
EBUS-guided cryobiopsy of mediastinal and hilar lymph nodes has shown to be a useful diagnostic tool to obtain tissue for histological analysis and further targeted therapies in lung malignancies. Due to the large size and better quality of the tissue samples, a higher diagnostic yield than with transbronchial needle aspiration (TBNA) can be expected, especially in non-solid tumors. In previous studies different biopsy protocols were used. The freezing time of cryoprobe (which defines the sample sizes) ranged from 3 to 7 s and the number of biopsies was between 1 and 4 samples. It is therefore unclear what freezing times and biopsy frequency are required to obtain the best histological information. This study will analyze whether the freezing time influences the diagnostic yield in CB of mediastinal lymphadenopathies. Additionally we will evaluate the influence of the number of biopsies on the diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* At least one mediastinal lesion or hilar 1 cm or longer in the short axis requiring diagnostic bronchoscopy
* Age between 18 and 90 years
* Written informed consent after participant's information

Exclusion Criteria:

* Age < 18 and > 90 years
* Lacking ability to form an informed consent (including impaired judgement, communication barriers)
* Contraindication against bronchoscopy (e.g. co-morbidities)
* Mediastinal abscess or cyst
* Extraordinary blood supply of the lesion visualized by EBUS bronchoscope
* INR > 1.5 or Thrombocytes < 100 G/l
* Clopidogrel or other new antiplatelet drugs within 7 days before biopsy (salicylic acid alone allowed)
* Anticoagulation with NOAC within 48 hours before biopsy
* Pulmonary lesions suspicious of lung carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | from date of randomization to the time of the first documented results, assessed up to 100 weeks
  Primary outcome measure is diagnostic yield according to the ATS consensus 2024 of EBUS-guided CB using two different freezing times (3sec./6.sec.).

SECONDARY OUTCOMES:
overall rate of suitability for histopathological examination | from the date of randomization to the time of the first documented results, assessed up to 100 weeks
the size of the harvested tissue (mm2) | from date of randomization to the time of the first documented results, assessed up to 100 months
), isolated and cumulative diagnostic yield of the first, second, third and fourth cryobiopsy | from date of randomization to the time of the first documented results, assessed up to100 weeks
time of the procedure | from the date of randomization to the time of the first documented results, assessed up to 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jürgen Hetzel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fan Y, Zhang AM, Wu XL, Huang ZS, Kontogianni K, Sun K, Fu WL, Wu N, Kuebler WM, Herth FJF. Transbronchial needle aspiration combined with cryobiopsy in the diagnosis of mediastinal diseases: a multicentre, open-label, randomised trial. Lancet Respir Med. 2023 Mar;11(3):256-264. doi: 10.1016/S2213-2600(22)00392-7. Epub 2022 Oct 22. PMID 36279880
- [Background] Zhang J, Guo JR, Huang ZS, Fu WL, Wu XL, Wu N, Kuebler WM, Herth FJF, Fan Y. Transbronchial mediastinal cryobiopsy in the diagnosis of mediastinal lesions: a randomised trial. Eur Respir J. 2021 Dec 9;58(6):2100055. doi: 10.1183/13993003.00055-2021. Print 2021 Dec. PMID 33958432